CLINICAL TRIAL: NCT06996054
Title: DEVELOPMENT AND EVALUATION OF A MULTIFACETED SCHOOL-BASED INTERVENTION TO PROTECT MENTAL HEALTH AND PREVENT SUICIDAL BEHAVIOR AMONG ADOLESCENTS IN SPAIN
Brief Title: Effects of a Multifaceted School-Based Intervention to Protect Mental Health and Prevent Suicidal Behaviour in Adolescents in Spain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació d'investigació Sanitària de les Illes Balears (Other Government)
Collaborators: University of the Balearic Islands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AP-15017/2024
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Suicide Attempt; Depression; Adolescent Mental Health; Self-Harm; Suicidal Ideation and Behavior
Keywords: School-based intervention; Suicide prevention; Suicidal ideation; Suicidal behavior; Depression; Adolescents; Mental health promotion; Psychoeducation; Gatekeeper training; Teachers; Parents; Digital health; Cluster randomized controlled trial; Spain; Secondary education; Emotional regulation; Self-harm
MeSH Terms: conditions — Suicide, Attempted; Depression; Self-Injurious Behavior; Suicidal Ideation; Behavior; Suicide Prevention; Emotional Regulation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional study (Experimental): Participants in this group will receive a multifaceted school-based intervention designed to prevent suicidal behavior and promote mental health. The intervention includes:
  * Psychoeducational sessions for students: Four weekly classroom-based sessions (90 minutes each), led by trained psychologists. Topics include mental health literacy, emotional regulation, identification of suicide risk, and help-seeking skills.
  * Digital co-intervention for parents and teachers: Access to a web-based platform delivering four multimedia modules with videos, podcasts, and educational content to improve suicide-related knowledge, self-efficacy, and referral practices.
  Interventions: Behavioral: Multifaceted School-Based Mental Health and Suicide Prevention Program
- Control (No Intervention): Participants in this group will receive a minimal intervention consisting of educational posters about mental health and suicide prevention displayed in classrooms. No additional training or sessions will be provided to students, parents, or teachers.

INTERVENTIONS:
Behavioral: Multifaceted School-Based Mental Health and Suicide Prevention Program — Pupils will receive a four-session psychoeducational programme, delivered weekly by trained psychologists during school hours, covering mental health literacy, emotion regulation, identification of suicide risk, and help-seeking skills. Concurrently, parents and teachers will access a digital co-intervention through a custom-designed platform with four multimedia modules.
  Arms: Interventional study

SUMMARY:
What is this study about? This study aims to find out if a school-based program can help improve mental health and prevent suicidal thoughts and behaviors in teenagers in Spain. Suicide is one of the leading causes of death among young people. Many teens who think about or attempt suicide are also struggling with mental health problems like depression. Schools offer a unique opportunity to help because almost all adolescents attend school regularly.

What will happen in the study?

The study will include about 2,280 students aged 12 to 16 years from 38 secondary schools in the Balearic Islands, Spain. Schools will be randomly assigned to one of two groups:

Intervention group: Students will participate in four weekly classroom sessions led by trained psychologists. These sessions will help students learn about mental health, manage their emotions, recognize signs of distress in themselves or others, and ask for help when needed. At the same time, parents and teachers will follow a digital training program with videos and resources to help them support students' mental health and recognize warning signs.

Control group: Students will receive a minimal intervention, which includes educational posters displayed in classrooms.

What is the purpose of this program? The main goal is to reduce suicidal thoughts and behaviors. The program also aims to improve students' overall mental well-being, reduce depression symptoms, and encourage help-seeking behaviors. It also helps parents and teachers feel more confident in supporting teens who may be at risk.

How will the study be evaluated? Students will complete questionnaires at the start of the study and again after six months. These surveys will ask about mental health, suicidal thoughts, emotional well-being, self-harm, substance use, and experiences with bullying. Parents and teachers will also complete surveys about their knowledge and confidence in supporting students.

Why is this study important? There is an urgent need to find effective ways to prevent suicide and support young people's mental health. This program involves students, families, and schools in working together to create a safe and supportive environment. If the program works, it could be used in schools throughout Spain and possibly in other countries too.

Who is funding this study? The study is funded by Fundación Mutua Madrileña.

DETAILED DESCRIPTION:
Background Adolescent suicide is a critical public health concern and one of the leading causes of death among youth globally. In Spain, suicide has been the primary external cause of death since 2008. Rates are especially concerning among adolescents and young adults. Depression and other mental health disorders are major risk factors associated with suicidal thoughts and behaviors in this population.

Schools provide a strategic setting for suicide prevention and mental health promotion, as they offer direct and repeated access to adolescents during a critical stage of emotional development. The involvement of teachers and families is also crucial, as they play a key role in identifying and supporting students at risk.

This study is a two-arm, cluster-randomised controlled trial designed to evaluate the effectiveness of a multifaceted school-based intervention to reduce suicidal ideation and behavior and promote mental health in adolescents aged 12 to 16 years. A total of 38 secondary schools in the Balearic Islands, Spain, will be randomly allocated in a 1:1 ratio to either the intervention or control group, with 2,280 students expected to participate.

Intervention Description

The intervention comprises two components:

1. Student-focused psychoeducational program: Delivered by trained psychologists in four weekly classroom sessions (90 minutes each), this component is based on a comprehensive model of suicide prevention and mental health promotion. The sessions include:

   * Mental health literacy and stigma reduction
   * Emotional regulation and coping strategies
   * Recognition of warning signs and crisis response
   * Promotion of help-seeking behavior and strengthening of social support networks Sessions incorporate dynamic group activities to enhance engagement and learning. The program is designed to foster a safe environment for sharing and reflection.
2. Digital co-intervention for parents and teachers: Delivered through a custom-built digital platform, this component includes four knowledge modules with videos, podcasts, and additional educational resources. The content aligns with the student sessions and aims to improve suicide-related knowledge, reduce stigma, increase self-efficacy, and support identification and referral of at-risk students. Access to the platform is monitored through user self-reports and automated engagement tracking.

The control group will receive a minimal intervention in the form of educational posters on mental health and suicide prevention placed in classrooms.

Outcomes and Data Collection Primary and secondary outcomes will be assessed using validated instruments at baseline and six-month follow-up. Primary outcomes include suicidal ideation and behavior. Secondary outcomes include symptoms of depression, psychological well-being, self-harm, substance use, internet addiction, bullying, and help-seeking behaviors. Teachers and parents will report on suicide-related knowledge, self-efficacy, and student referrals.

Process evaluation will be conducted through qualitative interviews with a subsample of students, parents, and teachers to assess the implementation, acceptability, and perceived impact of the intervention.

Data will be analyzed using generalized linear mixed models to account for the clustering of students within schools. Multiple imputation will be used to address missing data. The primary analysis will follow an intention-to-treat approach.

Significance This study addresses a critical gap in the evidence base for suicide prevention programs in Spain. It aims to provide robust data on the effectiveness of a scalable, cost-effective, and digitally enhanced intervention. If successful, the intervention may support wider implementation in schools and contribute to improved mental health outcomes and suicide prevention strategies at the national level.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in the 2nd or 3rd year of compulsory secondary education during the 2026-2027 academic year in the Balearic Islands, Spain.
* Aged between 12 and 16 years at the time of recruitment.
* Provision of written informed consent from both the student and at least one parent/legal guardian.
* Attending school centres with a student population composed of no more than 75% of a single gender.
* Enrollment in a participating classroom randomly selected for the study.

Exclusion Criteria:

* Presence of cognitive, developmental, or language impairments that, in the judgment of school staff or study personnel, would prevent the student from understanding the intervention content or completing the study assessments reliably.
* Students currently receiving intensive psychological or psychiatric treatment for acute suicidality or severe mental health conditions that require individualized clinical management beyond the scope of a school-based programme.
* Students or parents who explicitly decline participation in specific intervention components, such as group discussions on suicide or mental health.
* Participation in a concurrent school-based mental health programme that could confound the effects of the intervention.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2280 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Severity of Suicidal Ideation | Baseline and 6-month follow-up
  Change in the severity of suicidal ideation as assessed by the Spanish version of the Suicidal Paykel Scale. This 5-item scale evaluates the presence and intensity of suicidal thoughts over the previous year. Responses are dichotomous (Yes/No) and produce a score ranging from 0 (no ideation) to 5 (high severity). A higher total score indicates greater suicidal ideation severity.

SECONDARY OUTCOMES:
Suicide Attempts | Baseline and 6-month follow-up
  Proportion of students reporting a suicide attempt in the past year, assessed through item 5 of the Suicidal Paykel Scale ("Have you ever tried to end your life?").
Depressive Symptoms | Baseline and 6-month follow-up
  Severity of depressive symptoms measured using the Spanish version of the Beck Depression Inventory-II (BDI-II), a 21-item questionnaire. Scores range from 0 to 63, with higher scores indicating greater symptom severity.
Well-being | Baseline and 6-month follow-up
  Subjective well-being measured using the Spanish version of the WHO-5 Well-Being Index, a 5-item scale with scores ranging from 0 (worst) to 25 (best).
Self-Harm | Baseline and 6-month follow-up
  Incidence and characteristics of self-injury behaviors assessed using the 15-item Spanish version of the Self-Harm Questionnaire (DSHI). Includes method, frequency, motivation, and context of self-harm.
Internet Addiction | Baseline and 6-month follow-up
  Problematic internet use assessed using the Spanish version of the Internet Addiction Test (IAT), a 20-item measure with scores from 20 to 100.
Substance Use | Baseline and 6-month follow-up
  Risk of substance use disorder measured using the Spanish version of the CRAFFT Screening Test. Scores range from 0 to 6; scores ≥2 indicate high risk.
Bullying Involvement | Baseline and 6-month follow-up
  Bullying experiences assessed via the Bull-S Test, which includes peer and teacher nominations to identify victims and aggressors within the classroom.
Help-Seeking Behaviors | Baseline and 6-month follow-up
  Student-reported intentions and behaviors related to seeking help for mental health issues, collected through study-specific questionnaires.

OTHER OUTCOMES:
Gatekeeper Knowledge of Suicide (Teachers and Parents) | Pre- and post-intervention (6 months)
  Knowledge of suicide risk factors and appropriate intervention strategies among parents and teachers, assessed using a study-specific questionnaire aligned with digital module content.
Gatekeeper Self-Efficacy in Suicide Risk Intervention | Pre- and post-intervention (6 months)
  Self-perceived efficacy in identifying and intervening with students at risk of suicide, measured via a 5-item Likert-scale questionnaire.

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in published articles will be shared after de-identification. This includes data for all primary and secondary outcome measures (e.g., suicidal ideation, depression scores, self-harm, internet addiction, bullying involvement, and well-being), as well as demographic variables (e.g., age, sex, school characteristics).
  Data will be shared in a de-identified format to protect participant confidentiality. No data that could directly identify participants will be shared. Data will be made available to qualified researchers whose proposed use of the data has been approved by an independent review committee and who agree to sign a data access agreement.
  Data will be available beginning 12 months after publication of the main results and will remain available for 5 years.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available beginning 12 months after publication of the main results and will remain available for 5 years.
Access Criteria: De-identified individual participant data (IPD) and supporting documentation (e.g., study protocol, statistical analysis plan) will be made available to qualified researchers affiliated with academic institutions, non-profit organizations, or public health agencies.
  Researchers must submit a methodologically sound proposal outlining the purpose of the analysis, data requirements, and plans for ethical data use. Access will be granted upon approval by an independent review committee.
  Researchers will be required to sign a data use agreement that includes commitments to:
  * Use the data only for the approved purpose;
  * Not attempt to re-identify participants;
  * Maintain data confidentiality and security.
  * Approved users will receive access to the data through a secure, password-protected data repository managed by the study sponsor or affiliated institution.